CLINICAL TRIAL: NCT02542475
Title: Low Field Magnetic Stimulation: Open Label Study.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Michael Rohan, Imaging Physicist, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001011
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Mood Disorders; Anxiety
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mood Improvement (Experimental): Mood change with daily Low Field Magnetic Stimulation in participants suffering from affective disorders and/or anxiety
  Interventions: Device: Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Low Field Magnetic Stimulation — The Low Field Magnetic Stimulation (LFMS) procedure is an application of a series of electromagnetic pulses to the brain. The field and timing parameters of the LFMS pulses, such as pulse timing, duration, frequency, and electric and magnetic field distribution and direction are different from other neurostimulation methods. LFMS electromagnetic fields are significantly weaker (< 100x) than those used in ECT and rTMS.
  Other Names: LFMS

SUMMARY:
To assess the effects of daily LFMS treatments for those suffering from affective or anxiety symptoms. We hypothesize a reduction in affective and or anxiety symptoms after active treatment over the period of one week, with improvement through the following week.

DETAILED DESCRIPTION:
The Low Field Magnetic Stimulation (LFMS) procedure is an application of a series of electromagnetic pulses to the brain. The field and timing parameters of the LFMS pulses, such as pulse timing, duration, frequency, and electric and magnetic field distribution and direction are different from other neurostimulation methods. LFMS electromagnetic fields are significantly weaker (< 100x) than those used in ECT and rTMS.

LFMS was discovered at McLean Hospital and has thus far been studied as an experimental antidepressant treatment at McLean Hospital. LFMS is also being studied at Massachusetts General Hospital and 5 other hospitals in an NIH sponsored trial (RAPID) as well as in studies at Cornell-Weill School of Medicine. The mechanism of action for the antidepressant effects of LFMS is hypothesized to be an interaction between the electromagnetic fields and neurons in cortical regions, brought about by low level electrical stimulation applied with particular timing.

The current study proposes to assess the effects of daily LFMS treatments in participants suffering from affective disorders and/or anxiety. This is an open-label study. All subjects will receive active LFMS treatments. Potential subjects will be referred to the study by their clinicians and will be pre-screened by phone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be accepted into the study upon written referral by a McLean clinician or outside psychiatrist.
2. Subjects will be men or women over the age of 18.
3. Subjects must have failed at least one FDA approved treatment before enrolling in this study.
4. Subjects must be capable of providing informed consent.
5. Subjects must have either a Hamilton Depression Rating Scale (HDRS) score > 14 indicating moderate depression or Hamilton Anxiety Rating Scale (HARS) score > 18 indicating moderate anxiety.

Exclusion Criteria:

1. Dangerous or active suicidal ideation.
2. Pregnant or planning on becoming pregnant.
3. Recent history (within 3 days) of ECT or TMS treatment.
4. Substance abuse (cannot meet DSM criteria for substance abuse, no significant drug abuse within last 3 months, no history of dependence in last year, no drug use within last month, other than marijuana use).
5. Current psychosis.
6. Contraindications for MRI: Presence of a pacemaker, neurostimulator, or metal in head or neck.
7. "Do Not Resuscitate" order in place (to avoid risk in the case of non-study-related accidents).

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Changes in daily mood after LFMS treatment using the Beck Depression Inventory (BDI) | 24 hrs
  Daily change in the BDI before and after each LFMS treatment
Change in mood after 5 days of LFMS treatment using the Hamilton Depression Rating Scale (HDRS) | 5 days
  Change in HDRS from before the first treatment to after the 5th (final) treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Rohan, Ph.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

REFERENCES:
- [Background] Rohan ML, Yamamoto RT, Ravichandran CT, Cayetano KR, Morales OG, Olson DP, Vitaliano G, Paul SM, Cohen BM. Rapid mood-elevating effects of low field magnetic stimulation in depression. Biol Psychiatry. 2014 Aug 1;76(3):186-93. doi: 10.1016/j.biopsych.2013.10.024. Epub 2013 Nov 12. PMID 24331545